CLINICAL TRIAL: NCT02033096
Title: A 4-Year Follow-up, Blinded-Outcomes Trial of Subjects Having Received Stannsoporfin or Placebo in Clinical Trial 64,185-202
Brief Title: Observational Follow-up of Participants From Clinical Trial 64,185-202 (NCT00850993)
Status: Completed | Type: Observational
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Other Study IDs: 64,185-203
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-08

CONDITIONS: Jaundice; Neonatal Hyperbilirubinemia
Keywords: stannsoporfin; hyperbilirubinemia; heme oxygenase
MeSH Terms: conditions — Jaundice; Hyperbilirubinemia, Neonatal; Hyperbilirubinemia | interventions — tin mesoporphyrin; Sodium Chloride; Phototherapy; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Cohort 1: Stannsoporfin 1.5 mg/kg: Cohort 1: Received one 1.5 mg/kg stannsoporfin injection (with phototherapy as needed) during participation in an earlier interventional trial (NCT00850993)
  Interventions: Drug: Stannsoporfin; Other: Phototherapy (as needed)
- Cohort 2: Stannsoporfin 3.0 mg/kg: Cohort 2: Received one 3.0 mg/kg stannsoporfin injection (with phototherapy as needed) during participation in an earlier interventional trial (NCT00850993)
  Interventions: Drug: Stannsoporfin; Other: Phototherapy (as needed)
- Cohort 3: Stannsoporfin 4.5 mg/kg: Cohort 3: Received one 4.5 mg/kg stannsoporfin injection (with phototherapy as needed) during participation in an earlier interventional trial (NCT00850993)
  Interventions: Drug: Stannsoporfin; Other: Phototherapy (as needed)
- Cohort 4: Placebo Control: Cohort 4: Received one sterile saline injection (with phototherapy as needed) during participation in an earlier interventional trial (NCT00850993)
  Interventions: Drug: Placebo Control; Other: Phototherapy (as needed)

INTERVENTIONS:
Drug: Stannsoporfin — No intervention was administered during this observational study
  Other Names: Experimental product
  Groups: Cohort 1: Stannsoporfin 1.5 mg/kg; Cohort 2: Stannsoporfin 3.0 mg/kg; Cohort 3: Stannsoporfin 4.5 mg/kg
Drug: Placebo Control — No intervention was administered during this observational study
  Other Names: Saline
  Groups: Cohort 4: Placebo Control
Other: Phototherapy (as needed) — No intervention was administered during this observational study
  Other Names: Standard Care

SUMMARY:
Observational follow-up of participants from earlier interventional trial 64,185-202 (NCT00850993).

No interventions were administered during this follow-up study.

ELIGIBILITY:
Inclusion Criteria:

Participants who received treatment in clinical trial 64,185-202 and for whom informed consent was given for long term safety followup

Exclusion Criteria:

Participants were excluded by the investigator for medical reasons or by parents/guardians withdrawing consent

Ages: 30 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies who participated in protocol 64,185-202 (NCT00850993)
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-10-20 (Actual); Primary Completion 2015-06-23 (Actual); Study Completion 2015-11-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | within 52 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Mallinckrodt

IPD SHARING:
Plan to Share IPD: No